CLINICAL TRIAL: NCT04922463
Title: PLASOMA Efficacy & Technology Health (PETH) Study: A Post-market Randomised Controlled Efficacy Study of PLASOMA on Wound Healing in Chronic Venous Leg Ulcers
Brief Title: PLASOMA Efficacy & Technology Health (PETH) Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The continuation of the study was rendered unreasonable due to the slow inclusion rate
Sponsor: Plasmacure (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PETH study
Record Dates: First submitted 2021-05-27; First posted 2021-06-10 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention)
- 1x PLASOMA (Experimental)
  Interventions: Device: PLASOMA
- 2x PLASOMA (Experimental)
  Interventions: Device: PLASOMA

INTERVENTIONS:
Device: PLASOMA — Treatment with cold plasma device
  Arms: 1x PLASOMA; 2x PLASOMA

SUMMARY:
This study is designed to examine beneficial effects of PLASOMA treatment compared to the standard of care on chronic venous leg ulcers (VLU) that match the size of the plasma area of the pad.

The intention is that the data obtained with this study will be used to:

1. Demonstrate comparative performance of PLASOMA (for two treatment frequencies)
2. Provide evidence for health technology assessments (HTA) of PLASOMA

DETAILED DESCRIPTION:
The PETH study will be an open label three-armed randomized controlled trial (RCT) on chronic VLU. The study will be performed at one study site in the Netherlands.

The three arms are:

* Control group: standard care for 12 weeks or until healing, whichever occurs first;
* Treatment group-1: standard care + PLASOMA treatment once per week for 12 weeks or until healing, whichever occurs first;
* Treatment group-2: standard care + PLASOMA treatment twice per week for 12 weeks or until healing, whichever occurs first.

After the treatment period there will be two follow up timepoints: 2 weeks after the end of the treatment period (FU1) and 12 weeks after the end of the treatment period (FU2).

Subjects will be allocated to one of the three arms according to a pre-defined randomization schedule.

Primary study parameters/outcome of the study:

Evaluate the percentage of wounds healed after 12 weeks of treatment with PLASOMA for two treatment frequencies: once per week and twice per week.

This will be done by comparing the treatment groups with the control group

ELIGIBILITY:
Inclusion criteria:

INCL1: have a slow-healing or non-healing lower leg ulcer presumed to be caused by venous insufficiency (VLU). The wound should have insufficient healing (<30% surface area reduction) during the last 2 weeks of standard wound care.

INCL2: have a wound with a minimum wound surface area of 0.5 cm2 and a maximum diameter of 6 cm (~28 cm2 wound surface area for circular wounds).

INCL3: have an Ankle Brachial Pressure Index (ABPI) between 0.8 and 1.3. Note 1: subject can be included based on a VLU diagnosis from anamnesis. Make sure an ABPI measurement is performed as soon as possible to verify the diagnosis. The subject has to be excluded if the ABPI is not between 0.8 and 1.3.

Note 2: For diabetic patients an ABPI measurement is not always reliable. Therefore, diabetic patients can be included based on a VLU diagnosis from anamnesis, but no ABPI measurement needs to be performed.

INCL4: have a minimum age of 18 years old.

INCL5: For home care treatments only: there is a grounded wall socket available for connection of PLASOMA.

Exclusion Criteria:

EXCL1: the subject has one or more of the following contraindications for PLASOMA:

* the wound is very exudative, i.e. wounds in which moisture is visible again within a few minutes after patting dry.
* any implanted active electronic device, such as a pacemaker, is present.
* an electronic medical device is attached to the body, including electronic life support equipment, hearing aids, glucose sensors and insulin pumps. If the sole purpose of the medical device is monitoring, the subject is not excluded, but it should be noted that use of PLASOMA together with such devices has not been tested and may lead to erroneous operation of the attached device during PLASOMA treatment.

Note: no exclusion if electronic medical device will be detached during PLASOMA treatment.

* a metal implant (including a stent) is present in the treatment area, i.e. the area between pad and electrode.
* a conductive connection from outside to inside the body at or near the heart is present, e.g. a catheter with electrolyte fluid.
* the subject has epilepsy
* the subject is pregnant

EXCL2: the subject uses systemic antibiotics.

EXCL3: the subject has any known malignant wound degeneration.

EXCL4: the subject receives treatment with immunosuppressive agents or oral corticosteroids; no exclusion if subject has received a stable dose for at least 2 months and the oral corticosteroid dose does not exceed 7.5 mg/day prednisone or equivalent.

EXCL5: the subject is receiving or likely to receive advanced wound dressings or advanced therapies- such as negative pressure therapy, hyperbaric oxygen therapy, biologicals (e.g. skin substitutes, growth factors), electrophysical therapy - for the to-be-treated wound.

EXCL6: the subject cannot (agree to) comply with the SOC.

EXCL7: the subject participates in another study which is likely to compromise the outcome of the PETH study or the feasibility of thesubject fulfilling the PETH study.

EXCL8: the subject is unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the percentage of wounds healed after 12 weeks of treatment with PLASOMA for two treatment frequencies: once per week and twice per week | 12 weeks

SECONDARY OUTCOMES:
Wound healing | 4 weeks
Time to healing | until 12 weeks
% Wounds with wound surface area reduction ≥50% | 4 weeks
Wound surface area reduction | 4 weeks
Wound surface area reduction | 12 weeks
Wound volume reduction | 4 weeks
Wound volume reduction | 12 weeks
Number of recurrences | 5 weeks
Number of recurrences | 9 weeks
Number of recurrences | 12 weeks
Scarring | FU1 (2 weeks after end of treatment)
Scarring | FU2 (12 weeks after end of treatment)
Quality of life - general | FU1 (2 weeks after end of treatment)
  RAND-36 questionnaire
Quality of life - wound specific | FU1 (2 weeks after end of treatment)
  Wound-QOL questionnaire
Wound pain | 20 weeks
  wound pain, using 0-10 numerical rating scale
Wound infection | until FU2 (12 weeks after end of treatment)
  wound infection (clinical classification)
Health Technology Assessment | 20 weeks
  resources used
Patient acceptability | 20 weeks
  subjects will be asked if they are happy with the PLASOMA treatment
Adverse Events with a potential relation to PLASOMA | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Koen Lim, Study Director — Plasmacure
Locations (2):
- Netherlands (2):
  - BBeterzorg, Sittard
  - Thebe Zorg Thuis, Tilburg

REFERENCES:
- [Result] Bakker O, Smits P, van Weersch C, Quaaden M, Bruls E, van Loon A, van der Kleij J. Improved Wound Healing by Direct Cold Atmospheric Plasma Once or Twice a Week: A Randomized Controlled Trial on Chronic Venous Leg Ulcers. Adv Wound Care (New Rochelle). 2025 Jan;14(1):1-13. doi: 10.1089/wound.2023.0196. Epub 2024 Jun 3. PMID 38687339